CLINICAL TRIAL: NCT00857272
Title: F38-27: An Evaluation of 2 Different Bowel Cleansing Preparations in Adult Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Braintree Laboratories (Industry)
Responsible Party: John McGowan, Associate Director, Clinical Research, Braintree Laboratories, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F38-27
Record Dates: First submitted 2009-03-05; First posted 2009-03-06 (Estimated); Results first posted 2010-09-28 (Estimated); Last update posted 2010-10-05 (Estimated); Status verified 2010-09

CONDITIONS: Colonoscopy
Keywords: colonoscopy; bowel preparation
MeSH Terms: interventions — Bisacodyl

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HalfLytely with 10mg bisacodyl (Active Comparator): Active control
  Interventions: Drug: PEG electrolyte lavage solution + bisacodyl
- HalfLytely with 5mg bisacodyl (Experimental): Investigational dose
  Interventions: Drug: PEG electrolyte lavage solution + bisacodyl - reformulation

INTERVENTIONS:
Drug: PEG electrolyte lavage solution + bisacodyl - reformulation — multi dose formulation (tablet/solution) for oral administration prior to colonoscopy
  Arms: HalfLytely with 5mg bisacodyl
Drug: PEG electrolyte lavage solution + bisacodyl — multi dose preparation (tablet/solution) for oral administration prior to colonoscopy
  Arms: HalfLytely with 10mg bisacodyl

SUMMARY:
To compare the safety and efficacy of 2 different bowel cleansing preparations prior to colonoscopy in adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female outpatients who are undergoing colonoscopy for a routinely accepted indications:
2. At least 18 years of age
3. Otherwise in good health, as determined by physical exam and medical history
4. If female, and of child-bearing potential, is using an acceptable form of birth control
5. Negative urine pregnancy test at screening, if applicable
6. In the Investigator's judgment, subject is mentally competent to provide informed consent to participate in the study

Exclusion Criteria:

1. Subjects with known or suspected ileus, gastrointestinal obstruction, gastric retention, bowel perforation, toxic colitis, or toxic megacolon
2. Subjects with impaired consciousness that predisposes them to pulmonary aspiration
3. Subjects who are undergoing colonoscopy for foreign body removal and decompression
4. Subjects with pre-existing electrolyte disturbances, such as dehydration, or those secondary to the use of diuretics
5. Subjects who are taking drugs that may affect electrolyte levels with the exception of routine diuretics
6. Subjects with known clinically significant electrolyte abnormalities such as hypernatremia, hyperphosphatemia, hypokalemia, or hypocalcemia
7. Subjects who are pregnant or lactating, or intending to become pregnant during the study
8. Subjects of childbearing potential who refuse a pregnancy test
9. Subjects who are allergic to any preparation components
10. Subjects who, in the opinion of the Investigator, should not be included in the study for any reason, including inability to follow study procedures
11. Subjects who have participated in an investigational clinical, surgical, drug, or device study within the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2009-02; Primary Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John McGowan, MPH, Study Director — Braintree Laboratories, Inc.
Locations (6):
- United States (6):
  - Advanced Clinical Research Institute, Anaheim, California
  - Advanced Clinical Research Institute, Orange, California
  - Medical Associates Research Group, San Diego, California
  - United Medical Research, New Smyrna Beach, Florida
  - Maryland Digestive Disease Research, Laurel, Maryland
  - Franklin Gastroenterology, Franklin, Tennessee

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HalfLytely With 5mg Bisacodyl | HalfLytely With 10mg Bisacodyl
Started | 154 (Includes 6 non-ITT patients that withdrew consent) | 154 (Includes 7 non-ITT patients that withdrew consent)
Completed | 145 | 145
Not Completed | 9 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HalfLytely With 5mg Bisacodyl | HalfLytely With 10mg Bisacodyl | Total
Number analyzed (Participants) | 154 | 154 | 308
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 110 | 116 | 226
  >=65 years | 44 | 38 | 82
Age Continuous [Mean (Standard Deviation); unit: years] | 56.8 (12.1) | 55.0 (13.0) | 55.9 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 90 | 168
  Male | 76 | 64 | 140
Region of Enrollment [Number; unit: participants]
  United States | 154 | 154 | 308

OUTCOME MEASURES:

1. Primary Outcome: Efficacy: Percentage of Patients With Successful Preparations Based on a 4 Point Scale
Description: Cleansing was scored with a four point scale used in previous bowel cleansing studies where 4 = "excellent" (no more than small bits of adherent feces/fluid); 3 = "good" (small amounts of feces or fluid not interfering with the exam); 2 = "fair" (enough feces or fluid to prevent a completely reliable exam); 1 = "poor" (large amounts of fecal residue requiring additional cleansing). For the primary efficacy endpoint (preparation success), grades of 4 and 3 were considered a "success" and grades of 2 or 1 were considered a "failure".
Time Frame: during colonoscopy
Population: The analysis population consists of patients that were randomized and took any portion of the study preparation and who did not discontinue prior to colonoscopy due to a reason of safety or efficacy.
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | HalfLytely With 5mg Bisacodyl | HalfLytely With 10mg Bisacodyl
Number analyzed (Participants) | 147 | 146
percent of participants | 77.6 [69.9 to 84.0] | 80.1 [72.7 to 86.3]
Statistical Analysis 1: Comparison: HalfLytely With 5mg Bisacodyl vs HalfLytely With 10mg Bisacodyl; The primary endpoint of preparation success was tested using a non-inferiority test based upon the difference D=P1-P2, Null Hypothesis H0: P1-P2<=D0 versus Alternative Hypothesis H1: P1-P2=D1>D0, Where P1 is the % of patients with successful preps in the HalfLytely 5mg group and P2 is the % of patients with successful preps in the HalfLytely 10mg group and D0 is the acceptable margin of equivalence equal to an absolute margin of 15%; Test type: Non-Inferiority or Equivalence — Fifteen percent has been established as an acceptable non-inferiority margin for evaluation of investigational bowel preparations in previous studies of FDA approved preparations (e.g. NuLytely, MoviPrep); p = 0.005, Chi-squared; Difference in success rates = -2.5, 95% CI 2-sided [-11.9 to 6.8]

ADVERSE EVENTS:
Arm/Group | HalfLytely With 5mg Bisacodyl | HalfLytely With 10mg Bisacodyl
Serious Adverse Events (participants affected / at risk) | 0/154 | 1/154
Other Adverse Events (participants affected / at risk) | 117/154 | 129/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HalfLytely With 5mg Bisacodyl (N=154) | HalfLytely With 10mg Bisacodyl (N=154)
urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
urosepsis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HalfLytely With 5mg Bisacodyl (N=154) | HalfLytely With 10mg Bisacodyl (N=154)
Overall Discomfort (General disorders) | 87 | 102 — Patient completed questionnaire - expected preparation symptoms were rated as "None", "Mild", "Bothersome", "Distressing" or "Severely Distressing"
Abdominal fullness (Gastrointestinal disorders) | 61 | 81 — Patient completed questionnaire - expected preparation symptoms were rated as "None", "Mild", "Bothersome", "Distressing" or "Severely Distressing"
Abdominal cramping (Gastrointestinal disorders) | 58 | 71 — Patient completed questionnaire - expected preparation symptoms were rated as "None", "Mild", "Bothersome", "Distressing" or "Severely Distressing"
Nausea (Gastrointestinal disorders) | 53 | 65 — Patient completed questionnaire - expected preparation symptoms were rated as "None", "Mild", "Bothersome", "Distressing" or "Severely Distressing"
Vomiting (Gastrointestinal disorders) | 15 | 10

LIMITATIONS AND CAVEATS:
Total number of patients experiencing a non-serious adverse event is based on all adverse events, not just those events above the reporting threshold of 3%

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 360 days from the time submitted to the sponsor for review. The sponsor cannot extend the embargo.